CLINICAL TRIAL: NCT05145504
Title: Evaluation of Biomarker IL-6 in Synovial Fluid in Obese and Normal Weight Patients Suffering From Gonarthrosis During Knee Arthroplasty Surgery.
Brief Title: Evaluation of IL-6 in Synovial Fluid in Obese and Normal Weight Patients Suffering From Gonarthrosis During PTA
Acronym: IL6PG
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: IL6PG
Record Dates: First submitted 2021-11-25; First posted 2021-12-06 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: IL-6 Concentration in the Synovial Fluid of Obese Patients is 100% Higher Than the IL-6 Concentration of the Synovial Fluid in Normal Weight Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 20 obese patients, with BMI ≥ 30
  Interventions: Diagnostic Test: Evaluation of IL-6 biomarkers in synovial fluid
- 20 normal weight patients with BMI between 18.5 - 24.9 inclusive
  Interventions: Diagnostic Test: Evaluation of IL-6 biomarkers in synovial fluid

INTERVENTIONS:
Diagnostic Test: Evaluation of IL-6 biomarkers in synovial fluid — Evaluation of IL-6 biomarkers in synovial fluid in obese and normal weight patients with gonarthrosis

SUMMARY:
Evaluate the concentration of IL-6 in the synovial fluid of obese patients suffering from gonarthrosis during knee arthroplasty surgery

ELIGIBILITY:
Inclusion Criteria:

* age between 55 and 85 years inclusive,
* Normal weight patients with BMI 18-24.9 included
* Obese patients with BMI ≥ 30
* Patients suffering from gonarthrosis awaiting knee arthroplasty surgery
* Patients awaiting knee replacement surgery
* Patients who agree to sign informed consent

Exclusion Criteria:

* Patients under 55 years of age.
* Patients over 85 years of age
* Patients suffering from diabetes mellitus
* Patients who are unable to understand
* Patients with severe neurological disorders or severe disability
* Rheumatoid arthritis patients
* Cancer patients
* Patients on immunosuppressive therapy

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is made up of obese and normal weight patients, of age, undergoing knee replacement surgery for gonarthrosis
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Evaluate whether the IL-6 concentration in the synovial fluid of obese patients is 100% higher than the IL-6 concentration of the synovial fluid in normal weight patients | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy